CLINICAL TRIAL: NCT02276495
Title: Does Single Injection Adductor Canal Block Improve Postoperative Analgesia in Patients Receiving Periarticular Local Anesthesia Injections for Total Knee Arthroplasty?
Brief Title: Can Single-Injection Adductor Canal Blocks Improve PostOp Pain Relief in Patients Undergoing Total Knee Arthroplasty?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Joseph Brian Rinehart, Assistant Clinical Professor, University of California, Irvine
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20141217; UCIANES06 (Other: UCIANE)
Record Dates: First submitted 2014-10-20; First posted 2014-10-28 (Estimated); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Pain Management
Keywords: pain management for total knee arthroplasty
MeSH Terms: conditions — Agnosia | interventions — Sodium Chloride; Ropivacaine; Epinephrine; Ketorolac; Clonidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ACB Control + Local Infiltration (Experimental): ACB Control - 20 ml saline injection for ACB + Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline
  Interventions: Other: ACB Control - 20 ml saline injection for ACB; Drug: Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline
- ACB Study + Local infiltration (Experimental): ACB Study - 20 ml 0.5% Ropivacaine for Adductor Canal Block + Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline
  Interventions: Drug: ACB Study - 20 ml 0.5% Ropivacaine for Adductor Canal Block; Drug: Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline
- ACB Study Only (Experimental): ACB Study - 20 ml 0.5% Ropivacaine for Adductor Canal Block
  Interventions: Drug: ACB Study - 20 ml 0.5% Ropivacaine for Adductor Canal Block

INTERVENTIONS:
Other: ACB Control - 20 ml saline injection for ACB — Adductor Canal Block Control (20 ml saline injection)
  Arms: ACB Control + Local Infiltration
Drug: ACB Study - 20 ml 0.5% Ropivacaine for Adductor Canal Block — Adductor Canal Block Study (20 ml 0.5% Ropivacaine)
  Arms: ACB Study + Local infiltration; ACB Study Only
Drug: Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline — 100 mLs of a solution containing:
  Ropivacaine 2 mg/mL (49.25 mL) + Epinephrine 1 mg/mL (0.5 mL) + Ketorolac 30mg/mL (1mL) + Clonidine 100 mcg/mL (0.8 mL) + 0.9% Normal saline (48.45 mL)
  Arms: ACB Control + Local Infiltration; ACB Study + Local infiltration

SUMMARY:
The purpose of the study is to determine the effect of a single injection adductor canal block (ACB) on pain scores within 24 hours post total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA), also known as total knee replacement, has been associated with a significant pain burden in the postoperative period. Methods to manage pain associated with this operation have in the past included injecting pain medication into the epidural space of the spinal cord, around a peripheral nerve, around the space surrounding the joint, or a combination of pain management techniques.

In recent years, the femoral nerve block (injection of pain medication around the peripheral nerve, specifically the femoral nerve) has been proposed as an effective way to manage pain while sparing many of the undesirable side effects of narcotic pain medications. Traditional techniques of the femoral nerve block involve the injection of pain medication around the peripheral nerve at the level of the groin area. A nerve block at this point in the path of the femoral nerve affects all of the musculature of the front part of the thigh as well as the nerves responsible for sensation to the majority of the knee joint. The femoral nerve block performed at the level of the groin provides an excellent level of pain relief at the knee joint, but is also associated with weakness of the quadriceps muscle. The resultant quadriceps weakness can both slow the physical therapy process and be a risk factor for post-operative falls. Participation in physical therapy is a critical component of the rehabilitation process and is started as soon as tolerated by the patient. The ideal pain management technique would provide the same degree of pain relief as the femoral nerve block while preserving the strength in the front part of the thigh muscles.

One suggested technique to achieve both of these goals is the injection of a large volume dilute local pain medication mixture around the joint during surgery. This has been used as a substitute to provide pain relief around the joint while maintaining strength in the quadriceps muscle and the ability to participate in physical therapy. This technique however, does not last long since the medication disperses away from the joint space.

A variation of the femoral nerve block in the lower thigh, within a space called the adductor canal, has been demonstrated to provide equivalent amounts of pain relief as a proximal femoral nerve block along with preservation of motor function to the quadriceps muscle. What is not as well-established is whether the combination of injecting pain medication directly around the joint space in the knee along with a single injection of pain medication in the adductor canal in the lower thigh can improve pain scores and extend the duration of pain relief provided compared to only an injection around the joint space.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age 18+ years old having total knee arthroplasty (TKA) at UCI Medical Center
* American Society of Anesthesiologists physical status I to III

Exclusion Criteria:

* Allergy to local anesthetics
* Pregnancy
* Nursing Mothers
* Children <18 years of age
* Renal impairment (GFR<60 mL/min/1.73m2)
* Hepatic Impairment (active hepatitis, elevated AST or ALT, jaundice)
* Opioid tolerant patients (defined as greater than 30 mg Morphine equivalent consumed daily)
* Patients that are diabetic with peripheral neuropathy
* BMI greater than 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rinehart, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Background] Wylde V, Rooker J, Halliday L, Blom A. Acute postoperative pain at rest after hip and knee arthroplasty: severity, sensory qualities and impact on sleep. Orthop Traumatol Surg Res. 2011 Apr;97(2):139-44. doi: 10.1016/j.otsr.2010.12.003. Epub 2011 Mar 8. PMID 21388906
- [Background] Robbins SM, Rastogi R, McLaughlin TL. Predicting acute recovery of physical function following total knee joint arthroplasty. J Arthroplasty. 2014 Feb;29(2):299-303. doi: 10.1016/j.arth.2013.06.033. Epub 2013 Jul 26. PMID 23891055
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Buvanendran A, Kroin JS. Multimodal analgesia for controlling acute postoperative pain. Curr Opin Anaesthesiol. 2009 Oct;22(5):588-93. doi: 10.1097/ACO.0b013e328330373a. PMID 19606021
- [Background] Paul JE, Arya A, Hurlburt L, Cheng J, Thabane L, Tidy A, Murthy Y. Femoral nerve block improves analgesia outcomes after total knee arthroplasty: a meta-analysis of randomized controlled trials. Anesthesiology. 2010 Nov;113(5):1144-62. doi: 10.1097/ALN.0b013e3181f4b18. PMID 20966667
- [Background] Feibel RJ, Dervin GF, Kim PR, Beaule PE. Major complications associated with femoral nerve catheters for knee arthroplasty: a word of caution. J Arthroplasty. 2009 Sep;24(6 Suppl):132-7. doi: 10.1016/j.arth.2009.04.008. Epub 2009 Jun 24. PMID 19553071
- [Background] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Background] Mudumbai SC, Kim TE, Howard SK, Workman JJ, Giori N, Woolson S, Ganaway T, King R, Mariano ER. Continuous adductor canal blocks are superior to continuous femoral nerve blocks in promoting early ambulation after TKA. Clin Orthop Relat Res. 2014 May;472(5):1377-83. doi: 10.1007/s11999-013-3197-y. PMID 23897505
- [Background] Ng FY, Ng JK, Chiu KY, Yan CH, Chan CW. Multimodal periarticular injection vs continuous femoral nerve block after total knee arthroplasty: a prospective, crossover, randomized clinical trial. J Arthroplasty. 2012 Jun;27(6):1234-8. doi: 10.1016/j.arth.2011.12.021. Epub 2012 Feb 8. PMID 22325963
- [Background] Teng Y, Jiang J, Chen S, Zhao L, Cui Z, Khan MS, Du W, Gao X, Wang J, Xia Y. Periarticular multimodal drug injection in total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1949-57. doi: 10.1007/s00167-013-2566-0. Epub 2013 Jun 20. PMID 23783531

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the main operating room from January 2015 through December of 2019. Recruitment was prolonged due to PI changes secondary to personnel leaving the university.
Groups:
- Joint Infiltration Only: ACB Control - 20 ml saline injection for ACB + Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline
  ACB Control - 20 ml saline injection for ACB: Adductor Canal Block Control (20 ml saline injection)
  Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline: 100 mLs of a solution containing:
  Ropivacaine 2 mg/mL (49.25 mL) + Epinephrine 1 mg/mL (0.5 mL) + Ketorolac 30mg/mL (1mL) + Clonidine 100 mcg/mL (0.8 mL) + 0.9% Normal saline (48.45 mL)
- ACB + Joint Infiltration: ACB Study - 20 ml 0.5% Ropivacaine for Adductor Canal Block + Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline
  ACB Study - 20 ml 0.5% Ropivacaine for Adductor Canal Block: Adductor Canal Block Study (20 ml 0.5% Ropivacaine)
  Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline: 100 mLs of a solution containing:
  Ropivacaine 2 mg/mL (49.25 mL) + Epinephrine 1 mg/mL (0.5 mL) + Ketorolac 30mg/mL (1mL) + Clonidine 100 mcg/mL (0.8 mL) + 0.9% Normal saline (48.45 mL)
- ACB Only: ACB Study - 20 ml 0.5% Ropivacaine for Adductor Canal Block
  ACB Study - 20 ml 0.5% Ropivacaine for Adductor Canal Block: Adductor Canal Block Study (20 ml 0.5% Ropivacaine)
Period: Overall Study
Arm/Group | Joint Infiltration Only | ACB + Joint Infiltration | ACB Only
Started | 18 | 17 | 20
Completed | 18 | 17 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ACB Control + Local Infiltration: ACB Control - 20 ml saline injection for ACB + Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline
  ACB Control - 20 ml saline injection for ACB: Adductor Canal Block Control (20 ml saline injection)
  Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline: 100 mLs of a solution containing:
  Ropivacaine 2 mg/mL (49.25 mL) + Epinephrine 1 mg/mL (0.5 mL) + Ketorolac 30mg/mL (1mL) + Clonidine 100 mcg/mL (0.8 mL) + 0.9% Normal saline (48.45 mL)
- ACB Study + Local Infiltration: ACB Study - 20 ml 0.5% Ropivacaine for Adductor Canal Block + Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline
  ACB Study - 20 ml 0.5% Ropivacaine for Adductor Canal Block: Adductor Canal Block Study (20 ml 0.5% Ropivacaine)
  Local infiltration - 100 mLs of a solution containing: Ropivacaine + Epinephrine + Ketorolac + Clonidine + 0.9% Normal saline: 100 mLs of a solution containing:
  Ropivacaine 2 mg/mL (49.25 mL) + Epinephrine 1 mg/mL (0.5 mL) + Ketorolac 30mg/mL (1mL) + Clonidine 100 mcg/mL (0.8 mL) + 0.9% Normal saline (48.45 mL)
- Total: Total of all reporting groups
Arm/Group | ACB Control + Local Infiltration | ACB Study + Local Infiltration | ACB Study Only | Total
Number analyzed (Participants) | 18 | 17 | 20 | 55
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [60 to 74] | 68 [63 to 71] | 67 [62 to 76] | 67 [61 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 9 | 29
  Male | 7 | 8 | 11 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 17 | 20 | 55
Height (cm) [Median (Inter-Quartile Range); unit: centimeters] | 169 [160 to 179] | 167 [162 to 175] | 169 [156 to 175] | 169 [160 to 175]
Weight (lbs) [Median (Inter-Quartile Range); unit: pounds] | 198 [148 to 214] | 207 [170 to 219] | 181 [166 to 194] | 188 [154 to 214]

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: The primary outcome variable of interest is the median maximum pain score within 24 hours postoperative. Pain scores were rated on a scale from 0 - 10, with 0 being no discomfort/pain and 10 being worst imaginable pain.
Time Frame: within 24 hours postoperative
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Joint Infiltration Only | ACB + Joint Infiltration | ACB Only
Number analyzed (Participants) | 18 | 17 | 20
units on a scale | 5 [3.5 to 6] | 4.5 [2 to 5] | 4 [2 to 6]
Statistical Analysis 1: Comparison: Joint Infiltration Only vs ACB + Joint Infiltration vs ACB Only; Test type: Superiority; p = 0.668, Kruskal-Wallis

2. Secondary Outcome: Opioid Use
Description: 24 Hour post-surgical opioid use
Time Frame: within 24 hours postoperative
Measure: Median (Inter-Quartile Range); unit: Daily mg morphine equivalents
Arm/Group | Joint Infiltration Only | ACB + Joint Infiltration | ACB Only
Number analyzed (Participants) | 18 | 17 | 20
Daily mg morphine equivalents | 38 [18 to 66] | 0 [0 to 22] | 26 [0 to 45]
Statistical Analysis 1: Comparison: Joint Infiltration Only vs ACB + Joint Infiltration vs ACB Only; Test type: Superiority; p = 0.006, Kruskal-Wallis

3. Secondary Outcome: Ambulation Distance
Description: Total distance ambulated during physical therapy during first 24 hours
Time Frame: First 24 hours post-operative
Measure: Median (Inter-Quartile Range); unit: feet
Arm/Group | Joint Infiltration Only | ACB + Joint Infiltration | ACB Only
Number analyzed (Participants) | 18 | 17 | 20
feet | 140 [100 to 360] | 350 [225 to 370] | 95 [20 to 160]
Statistical Analysis 1: Comparison: Joint Infiltration Only vs ACB + Joint Infiltration vs ACB Only; Test type: Superiority; p = 0.013, Kruskal-Wallis

4. Other Pre Specified Outcome: Baseline Anxiety
Description: Self-reported subject anxiety prior to surgery
Time Frame: pre-operative day of surgery
Population: Data was incompletely collected across the study so no analysis performed
Arm/Group | Joint Infiltration Only | ACB + Joint Infiltration | ACB Only
Number analyzed (Participants) | 0 | 0 | 0

5. Other Pre Specified Outcome: Baseline Pain Score
Description: Baseline pain preoperatively
Time Frame: Preoperatively day of surgery
Population: Study data was incompletely collected across the study period so no analysis was performed
Arm/Group | Joint Infiltration Only | ACB + Joint Infiltration | ACB Only
Number analyzed (Participants) | 0 | 0 | 0

6. Other Pre Specified Outcome: NRS Pain Rating
Description: A modified pain score similar to VAS but rated from 0-10
Time Frame: Preop, PACU, and 4,8, 12, and 24 hours post-operatively.
Population: NRS scores were not collected during the study, so no analysis is performed.
Arm/Group | Joint Infiltration Only | ACB + Joint Infiltration | ACB Only
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All subjects were followed to 30 days post-operatively
Arm/Group | Joint Infiltration Only | ACB + Joint Infiltration | ACB Only
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/20

LIMITATIONS AND CAVEATS:
The PI changed twice during the study period, and the final PI left after the beginning of the COVID-19 pandemic. We have endeavored to collect as much of the original study data as possible in order to close out this record, but many measures were not collected (baseline anxiety & pain, NRS scores, etc). We have reported as much as possible based on hospital records and existing data that was collected during the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT02276495/Prot_SAP_000.pdf